CLINICAL TRIAL: NCT04398719
Title: Effect of Cannabidiol on Microglial Activation and Central Pain-Sensitization
Brief Title: CBD-Microglia PET Study
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Mohini Ranganathan, Associate Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2000026320
Record Dates: First submitted 2020-05-19; First posted 2020-05-21 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: CBD; Healthy
Keywords: Control; PET Scan; MRI Scan; Central Pain-Sensitization; Cannabidiol
MeSH Terms: interventions — (methyl-(11)C)N-acetyl-N-(2-methoxybenzyl)-2-phenoxy-5-pyridinamine; Magnetic Resonance Spectroscopy; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- CBD (Active Comparator)
  Interventions: Radiation: [11C]PBR28; Drug: Low-dose lipopolysaccharide; Drug: Intradermal Capsaicin
- Placebo (Placebo Comparator)
  Interventions: Radiation: [11C]PBR28; Drug: Low-dose lipopolysaccharide; Drug: Intradermal Capsaicin

INTERVENTIONS:
Radiation: [11C]PBR28 — The radiotracer, [11C]PBR28, will be administered at the beginning of each PET scan
  Other Names: PET scan
Drug: Low-dose lipopolysaccharide — Subjects will receive intravenous lipopolysaccharide.
  Other Names: LPS
Drug: Intradermal Capsaicin — A small dose of capsaicin will be administered by intradermal injection.

SUMMARY:
This study aims to examine the effect of cannabidiol (CBD) pre-treatment on brain microglial activation in healthy human subjects. Secondarily, this study aims to examine the effect of cannabidiol (CBD) pre-treatment on central pain-sensitization in healthy human subjects.

DETAILED DESCRIPTION:
This study aims to examine the effect of cannabidiol (CBD), pre-treatment, as Epidiolex, on brain microglial activation in healthy human subjects using [11C]PBR28 PET imaging. Secondarily, this study aims to examine the effect of cannabidiol (CBD) pre-treatment on central pain-sensitization in healthy human subjects. Lastly, this research study will also examine the relationship between brain microglial activation and central pain sensitization with CBD pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18- 55 years
2. No significant medical or neurological illness
3. No implanted metal devices that may pose a risk during MRI scanning
4. Within the annual permissible radiation exposure
5. Able to provide written informed consent.

Exclusion Criteria:

1. Current use of any medications
2. Presence of metal in the body
3. Pregnancy or lactation

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2021-05-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Microglial activation using [11C]PBR28 PET imaging | 10 Days
  Difference in microglial activation ([11C]PBR28 VT levels) between the 2 groups (e.g., CBD vs. placebo)

SECONDARY OUTCOMES:
Capsaicin-induced hyperalgesia | 10 Days
  Difference in capsaicin-induced hyperalgesia between the 2 groups (e.g., CBD vs. placebo)

CONTACTS AND LOCATIONS:
Overall Officials: Mohini Ranganathan, MD, Principal Investigator — Yale University
Locations (1):
- Connecticut Mental Health Center, New Haven, Connecticut, United States